CLINICAL TRIAL: NCT05089201
Title: A Pilot Study to Examine the Impact of a Therapy Dog Intervention on Loneliness and Related Health Outcomes in Vulnerable Populations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Waltham Petcare Science Institute (Unknown); Human Animal Bond Research Institute (HABRI) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: HM20021567
Record Dates: First submitted 2021-10-07; First posted 2021-10-22 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Loneliness; Depression; Anxiety; Quality of Life
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Animal-assisted interaction (AAI) (Experimental): Dogs and handlers will visit with patients for 20 minutes and discuss semi-scripted topics.
  Interventions: Behavioral: Animal-assisted interaction
- Conversational interaction (Active Comparator): Handlers will have a 20 minute semi-scripted conversation with patients.
  Interventions: Behavioral: Conversational control
- Treatment as usual (No Intervention): Patients will receive treatment as usual.

INTERVENTIONS:
Behavioral: Animal-assisted interaction — A dog-handler team or a handler alone will visit participants with a dog for approximately 20 minutes on 3 consecutive days during their inpatient hospital stay
  Arms: Animal-assisted interaction (AAI)
Behavioral: Conversational control — A handler alone will visit participants without a dog for approximately 20 minutes on 3 consecutive days during their inpatient hospital stay
  Arms: Conversational interaction

SUMMARY:
The purpose of this research study is to test whether an animal-assisted interaction (AAI) intervention is better than conversation with another person or treatment as usual for improving mood, anxiety, loneliness, quality of life, and indicators of health care services such as number of hospitalizations, length of hospital stay, and cost of services. Participants will be patients admitted for an inpatient stay at Virginia Commonwealth University Health who meet the study entry requirements.

DETAILED DESCRIPTION:
Participants will be randomly assigned (like the flip of a coin) to receive one of the following interventions:

1. Animal-assisted interaction (a dog-handler team will visit them in their hospital room)
2. Conversational interaction with just participants and the handler
3. Treatment as usual (the regular services patients are currently receiving in the hospital)

Participation in this study will last six months. This includes the three days on which participants will receive one of the interventions described above, plus completing some questionnaires online or by phone one month and six months after the baseline visit. These questionnaires will ask questions about pet ownership, relationship with pets participants have had, loneliness, depression, anxiety, health-related quality of life, significant life events in the past year, and social supports. Approximately 180 individuals will participate in this study.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Projected to be admitted to the hospital for the upcoming four days
* Speak English
* Able to provide consent.

Exclusion Criteria:

* Fear of, or allergy to, dogs
* Documented contact precautions
* Cognitive impairment that prevents consent or completion of measures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2021-11-16 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Number of participants enrolled | 2 years
  The number of eligible patients who sigh consent forms and are randomized to a condition
Attrition rate | 30 months
  Number of participants who do not complete the full study

SECONDARY OUTCOMES:
Change in loneliness | Baseline to 6 months
  Loneliness will be assessed using the 20-item Revised (Version 3) University of California, Los Angeles Loneliness Scale (Rev University of California, Los Angeles - Loneliness Scale).
Change in depression | Baseline to 6 months
  Depressive symptomology will be measured with the 10-item Center for Epidemiological Studies Depression short form (CESD-10) scale.
Change in anxiety | Baseline to 6 months
  Anxiety will be measured using the 20-item scale of the State-Trait Anxiety Inventory for Adults (STAI-AD).

CONTACTS AND LOCATIONS:
Overall Officials: Nancy R. Gee, PhD, Principal Investigator — Virginia Commonwealth University; Lisa Townsend, PhD, Study Director — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gee NR, Townsend L, Friedmann E, Barker SB, Thakre TP, Mueller MK. A pilot randomized controlled trial to examine the impact of a therapy dog intervention on loneliness in adult patients hospitalized in a psychiatric unit. Front Psychiatry. 2025 Dec 10;16:1582767. doi: 10.3389/fpsyt.2025.1582767. eCollection 2025. PMID 41450829
- [Derived] Gee NR, Townsend L, Friedmann E, Barker SB, Mueller MK. A Pilot Randomized Controlled Trial to Examine the Impact of a Therapy Dog Intervention on Loneliness in Hospitalized Older Adults. Innov Aging. 2024 Sep 16;8(11):igae085. doi: 10.1093/geroni/igae085. eCollection 2024. PMID 39790554